CLINICAL TRIAL: NCT00698490
Title: Study to Compare, in Healthy HSV Seronegative and HSV Seropositive Subjects, the Humoral and Cellular Immune Response of Herpes Simplex Candidate Vaccines Containing gD From Two Different Cell Lines and Using gD-Alum as Control
Brief Title: Humoral and Cellular Immune Response of Herpes Simplex (gD) Candidate Vaccines From 2 Different Cell Lines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208141/015
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Prophylaxis Herpes Simplex
Keywords: Herpes simplex; Herpes simplex candidate vaccine
MeSH Terms: conditions — Herpes Simplex

ARMS (5):
- Group A (Experimental): HSV-seronegative subjects
  Interventions: Biological: Adjuvanted herpes simplex (gD) candidate vaccine GSK 208141
- Group B (Experimental): HSV-seropositive subjects
  Interventions: Biological: Adjuvanted herpes simplex (gD) candidate vaccine GSK 208141
- Group C (Experimental): HSV-seronegative subjects
  Interventions: Biological: Adjuvanted herpes simplex (gD) candidate vaccine GSK 208141
- Group D (Experimental): HSV-seronegative subjects
  Interventions: Biological: Adjuvanted herpes simplex (gD) candidate vaccine GSK 208141
- Group E (Experimental): HSV-seronegative subjects
  Interventions: Biological: Herpes simplex virus containing gD-Alum

INTERVENTIONS:
Biological: Adjuvanted herpes simplex (gD) candidate vaccine GSK 208141 — Intramuscular injection, 3 doses, 2 different formulations
  Arms: Group A; Group B; Group C; Group D
Biological: Herpes simplex virus containing gD-Alum — Intramuscular injection, 3 doses
  Arms: Group E

SUMMARY:
The purpose of the study is to compare, in healthy HSV seronegative and HSV seropositive subjects, the humoral and cellular immune response of herpes simplex candidate vaccines containing gD from two different cell lines and using gD-Alum as control.

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years of age
* Written informed consent
* Female volunteers must be using contraception and should avoid becoming pregnant for the duration of the vaccination course
* Serology: Groups 1, 3, 4 and 5: HSV-1 AND HSV-2 seronegative (by gD2 ELISA); Group 2: HSV seropositive by gD2 ELISA before entry

Exclusion Criteria:

* Any previous vaccination against Herpes simplex.
* Any previous administration of MPL.
* Pregnancy or lactation.
* Patient is immuno-compromised or is receiving immuno-modifying therapy of any kind.
* Clinical signs of acute or febrile illness at the time of entry into the study.
* Any administration of immunoglobulins during the vaccination course or within one month of vaccination.
* Any vaccination within one week of study vaccination.
* Previous known hypersensitivity to vaccination or to any component of the vaccine.
* Simultaneous participation in any other clinical trial with an investigational drug or vaccine. Subjects currently in a follow-up period of a vaccine study can be included.
* Recent history of alcoholism or drug abuse (within the past 6 months).
* Life-threatening or serious cardiac (NYHA grades III-IV), gastrointestinal, hepatic, renal, hematological or immunological disorder which, in the opinion of the investigator, would preclude entry into the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 1995-08; Primary Completion 1997-01 (Actual); Study Completion 1997-01 (Actual)

PRIMARY OUTCOMES:
To evaluate in initially HSV-seronegative subjects the GMT's and the seroconversion rates of anti-gD2 antibodies (ELISA) | After the second and third doses of each vaccine
To evaluate in initially HSV-seronegative subjects, the GMT and the seropositivity rate of anti-HSV-2 neutralizing antibodies
To evaluate the cell-mediated immune (CMI) response (lymphoproliferation, secretion of interleukin 2 and γ interferon) | After the second and third dose of each vaccine formulation
To evaluate, in initially seronegative subjects and in initially seropositive subjects, the incidence and intensity of solicited local and general signs and symptoms | During 3 days after each dose of each vaccine
To evaluate in initially seropositive subjects, the GMT and the seropositivity rate of anti-gD2 antibodies (ELISA) and of anti-HSV-2 neutralizing antibodies | After 2 and 3 doses of vaccines

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Ghent, Belgium